CLINICAL TRIAL: NCT06228443
Title: A Single Dose, Randomized, Open-label, One-period Parallel Bioequivalence Study of Generic Leflunomide 20 mg Film-coated Tablets and Reference Product (Arava®) in Healthy Thai Male Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Generic Leflunomide 20 mg Film-coated Tablets and Reference Product Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Bio service (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BE23-031
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteer
Keywords: Leflunomide; Bioequivalence Study
MeSH Terms: interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leflunomide 20 mg Tablets (Test Drug) (Experimental): Leflunomide 20 mg Tablets ,1 x 20 mg, single dose fasting.
  Interventions: Drug: Leflunomide 20 mg Film-coated Tablet
- ARAVA® 20 mg Tablets (Reference Drug) (Active Comparator): ARAVA™ 20 mg Tablets,1 x 20 mg, single dose fasting.
  Interventions: Drug: ARAVA® 20 mg Film-coated Tablet

INTERVENTIONS:
Drug: Leflunomide 20 mg Film-coated Tablet — Leflunomide 20 mg Film-coated Tablet (Test Drug)
  Arms: Leflunomide 20 mg Tablets (Test Drug)
Drug: ARAVA® 20 mg Film-coated Tablet — ARAVA® 20 mg Tablets (Reference Drug)
  Other Names: Leflunomide 20 mg Film-coated Tablet
  Arms: ARAVA® 20 mg Tablets (Reference Drug)

SUMMARY:
This Study Aims to Assess the Relative Bioavailability, Including the Rate and Extent of Absorption, of 20 mg Leflunomide Tablets Compared to ARAVA® 20 mg Tablets. The Evaluation Will be Conducted Following a Single Oral Dose (1 x 20 mg Tablet) in Healthy Thai Male Volunteers Under Fasting Conditions.

DETAILED DESCRIPTION:
To compare the Bioavailability of leflunomide 20 mg tablets with that of ARAVA® 20mg tablets in healthy Thai Male Volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria

1. Healthy Thai male subjects between the ages of 18 to 55 years
2. Body mass index between 18.5 to 30.0 kg/m2.
3. Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening.

   Any abnormalities from the normal or reference range will be carefully considered clinically relevant by the physician as individual cases, documented in study files prior to enrolling the subject in this study
4. Male subjects who are not wishing to be a father of a child during the study or who are willing or able to use effective contraceptive e.g. condom or abstinence after check-in until 30 days after investigational product administration.
5. Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study

Exclusion Criteria

1. History of allergic reaction or hypersensitivity to leflunomide (especially previous Stevens-Johnson syndrome, toxic epidermal necrolysis or erythema multiforme), teriflunomide or any of the excipients in the tablet
2. History of allergic reaction or hypersensitivity to cholestyramine
3. History or evidence of clinically significant renal, hepatic, gastrointestinal, hematological (e.g. anemia), endocrine (e.g. hyper-/hypothyroid, diabetes), pulmonary or respiratory (e.g. asthma, COPD), cardiovascular (e.g. hyper-/hypotension), psychiatric, neurologic (e.g. convulsant), allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or any significant ongoing chronic medical illness
4. Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19
5. History about administration of COVID-19 vaccine within 30 days prior to check-in
6. History or evidence of easy bruising or bleeding, recurrent infections, fever, paleness or unusual tiredness
7. History or evidence of impairment of liver function
8. History or evidence of moderate to severe renal insuffici
9. History or evidence of severe hypoproteinaemia or nephrotic syndrome
10. Investigation with blood sample shows albumin level less than 3.5 g/dl or more than 5.2 g/dl at screening
11. Investigation with blood sample shows total protein level less than 6.6 g/dl or more than 8.7 g/dl at screening
12. History or evidence of severe immunodeficiency states
13. History or evidence of significantly impaired bone marrow function, significant anaemia, leucopenia or thrombocytopenia
14. Have sitting systolic blood pressure of less than 90 mmHg or more than 139 mmHg and diastolic blood pressure of less than 60 mmHg or more than 89 mmHg on screening day and check-in day. If abnormal blood pressure detects, the measurement should be repeated two more times after take a rest for at least 5 mins each. The last measurement value should be used to determine the subject's eligibility
15. History or evidence of colitis
16. History or evidence of peripheral neuropathy
17. History or evidence of galactose intolerance, the Lapp lactase deficiency or glucosegalactose malabsorption
18. History of problems with swallowing tablet or capsule
19. History of sensitivity to heparin or heparin-induced thrombocytopenia
20. Any condition possibly affecting drug absorption e.g. gastrectomy, enterectomy, gastritis or duodenal or gastric ulceration other than appendectomy
21. History of dehydration from diarrhea, vomiting, excess sweating or any other reason within 24 hours prior to check-in or prior to dosing
22. History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse (morphine, marijuana or methamphetamine)

23.12-lead ECG demonstrating QTc >450 msec, a QRS interval >120 msec or with an abnormality considered clinically significant at screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG will be repeated two more times and the average of the three QTc or QRS values will be used to determine the subject's eligibility.

24.Investigation with blood sample shows positive test for HBsAg

25.Abnormal liver function, ≥1.5 times of upper normal limit of reference range for ALT, AST or bilirubin levels at screening laboratory test

26.History or evidence of habitual use of tobacco or nicotine containing products and cannot abstain for at least 48 hours prior to check-in and continued for entire duration of the study

27.History or evidence of alcoholism or harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men and 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy, etc.)

28.History or eviden ce of alcohol consumption or alcohol-containing products and cannot abstain for at least 48 hours prior to check-in and continued for entire duration of the study or alcohol breath test shows positive result.In case of alcohol breath test result represents the alcohol concentration range of 1 - 10 mg% BAC and the physician carefully considers that the value came from other reasons, not from the alcohol drinking behavior of subjects, the test will be repeated two times separately, not more than 10 minutes. The result of the last time should be used for subject's eligibility which must be 0 mg%BAC.

29.History or evidence of habitual consume of tea, coffee, xanthine or caffeine containing products and cannot abstain for at least 48 hours prior to check-in and continued for entire duration of the study

30.Consume or drink juice of grapefruit or orange or pomelo or its supplement/containing products and cannot abstain for at least 7 days prior to check-in and continued for entire duration of the study

31.Use of prescription or nonprescription drugs (e.g. paracetamol, erythromycin, ketoconazole, cimetidine, DMARDs (e.g. methotrexate), coumarin anticoagulants (e.g. warfarin), indomethacin, ketoprofen, furosemide, ciprofloxacin, cefaclor, zidovudine, benzylpenicillin, repaglinide, pioglitazone, rosiglitazone, paclitaxel, rosuvastatin, etc.), herbal medications or supplements (e.g. St. John's wort), vitamins or mineral (e.g. iron) or dietary supplements within 14 days prior to check-in and continued for entire duration of the study

32.Participated in other clinical trials within 90 days prior to check-in (except for the subjects who drop out or withdrawn from the previous study prior to dosing) or still participates in the clinical trial or participates in other clinical trials during enrollment in this study

33.Blood donation or blood loss ≥ 1 unit (1 unit is equal to 350-450 mL of blood) within 90 days prior to check-in or during enrollment

34.Subjects with poor venous access or intolerant to venipuncture

35.Unwilling or unable to comply with schedule visit, treatment plan and other study procedures until end of study

36.Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that may impair the ability to provide written informed consent or cooperate with clinical team

37.Subjects who are employees of International Bio Service Co. Ltd. or Sponsor.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-04-26 (Estimated)

PRIMARY OUTCOMES:
Cmax | Blood samples collected over 72 hour period
  Maximum Observed Concentration - Metabolite A77 1726 in Plasma
AUC0-72 | Blood samples collected over 72 hour period
  Area Under the Concentration-time Curve From Time Zero to 72 Hours Post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Uthai Suvanakoot, Principal Investigator — International Bio service

IPD SHARING:
Plan to Share IPD: No